CLINICAL TRIAL: NCT04422743
Title: Effect of the Fixed Combination Citicoline 500 mg Plus Homotaurine 50 mg on Pattern Electroretinogram in Well Controlled Primary Open Angle Glaucoma: A Multicenter, Prospective, Randomized, Single Blind, Cross-over Study
Brief Title: Effect of Citicoline/Homotaurine on PERG in Primary Open Angle Glaucoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to covid 19 pandemy
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Gemma Caterina Maria Rossi, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NP2017
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2021-11

CONDITIONS: Glaucoma
Keywords: Pattern electroretinogram; visual field; quality of life; citicoline 500 mg plus homotaurine 50 mg
MeSH Terms: conditions — Glaucoma | interventions — Cytidine Diphosphate Choline; tramiprosate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard of care + citicoline plus homotaurine (CIT/HOMO) (Experimental): CIT/HOMO was supplemented for 4 months to the standard of care (SOC, i.e. topical intraocular pressure, IOP, lowering medication)
  Interventions: Dietary Supplement: Citicoline 500 mg plus Homotaurine 50 mg
- standard of care (No Intervention): only standard of care (SOC, i.e. topical IOP lowering medication) for 4 months

INTERVENTIONS:
Dietary Supplement: Citicoline 500 mg plus Homotaurine 50 mg — Citicoline 500 mg plus Homotaurine 50 mg was added to topical therapy
  Other Names: CIT/HOMO; Neuprozin®
  Arms: standard of care + citicoline plus homotaurine (CIT/HOMO)

SUMMARY:
the general purpose of the study is to evaluate the potential beneficial effects of supplementation of a fixed combination of Citicoline 500 mg plus Homotaurine 50 mg on retinal ganglion cells (RGCs) function in subjects with glaucoma by pattern electroretinogram.

DETAILED DESCRIPTION:
Secondary objectives are to assess effects on visual acuity, visual field changes, Quality of Life perception (NEI VFQ25 questionnaire), and safety (Incidence of adverse events)

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 75 years;
* diagnosis of primary OAG (POAG) from, at least, 3 years;
* visual acuity > 0.7 (7/10) decimals;
* refractive error < 5 D (spheric) and < 2D (toric);
* transparent diopter means (cornea and lens);
* controlled IOP (<18 mmHg, morning value) with beta-blockers and prostaglandin analogues as monotherapy or as associative therapy (fixed or unfixed);
* stable IOP<18 mmHg in the last 2 years;
* stable and unchanged topical therapy in the last 6 months;
* stable disease in the last 2 years (no more than -1 dB/year at MD of visual field);
* at least two reliable visual fields (Humphrey 24-2 Swedish interactive threshold algorithm -SITA- Standard) per year in the last 2 years;
* early to moderate visual field defect (MD <12 dB);
* electrophysiological (PERG) parameters alterations similar to glaucomatous pathology;
* written consent to participate to study procedures and data utilization in an anonymous form

Exclusion Criteria:

* ocular hypertension with normal optic nerve and visual field; angle closure glaucoma;
* congenital glaucoma; secondary glaucoma; normal tension glaucoma;
* history of recurrent uveitis/scleritis/herpes infection;
* pregnancy and breastfeeding;
* contraindication to Citicoline and/or Homotaurine
* contraindication to beta-blockers and prostaglandine analogues
* topical therapy with Brimonidine monotherapy or fixed combination (with timolol or brinzolamide)
* topical therapy with pilocarpine and aceclidine, monotherapy or fixed combination systemic or topical treatment with another neuroprotective agent in the last 4 months prior to enrollment
* systemic therapies affecting patients' performance in visual field examination (sedatives);
* glaucomatous scotomas within 10 degree from fixation
* any condition limiting the patient's ability to participate in the study;
* other ocular causes of visual field and PERG changes, such as cataract, myopic chorioretinopathy, macular diseases, retinal vascular occlusion, diabetic retinopathy;
* other systemic causes of visual field and PERG changes such as neurodegenerative disorders (Alzheimer's disease, Parkinson's disease, ALS, MS) or pituitary disorders;
* cerebral ischemia in the last 2 years
* any change in topical therapy in the 6 months prior to enrollment or during the study period concomitant participation to another clinical trial
* any previous filtering and/or retinal surgery;
* cataract surgery in the last 6 months;
* any previous laser treatment for glaucoma in the last 5 years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
To assess effects of adding the fixed combination of Citicoline 500 mg plus Homotaurine 50 mg (Neuprozin® - NP), one tablet a day, on PERG examination at four months of therapy, compared to standard of care alone, as add-on to standard therapy | 4 months of therapy 2 months of wash out 4 months without adding therapy
  changes in amplitude (microVolt)

SECONDARY OUTCOMES:
To assess effects of one tablet a day of the fixed combination of Citicoline 500 mg plus Homotaurine 50 mg (Neuprozin® - NP) on visual acuity | 4 months of therapy 2 months of wash out 4 months without adding therapy
  changes in visual acuity (decimals)
to assess effects of one tablet a day of the fixed combination of Citicoline 500 mg plus Homotaurine 50 mg (Neuprozin® - NP) on visual field | 4 months of therapy 2 months of wash out 4 months without adding therapy
  changes in mean deviation (deciBell-dB) and in pattern standard deviation (deciBell-dB) of visual field parameters
to assess effects of one tablet a day of the fixed combination of Citicoline 500 mg plus Homotaurine 50 mg (Neuprozin® - NP) on quality of life | 4 months of therapy 2 months of wash out 4 months without adding therapy
  changes in the total mean score and in the subscales of the 25 item National Eye Institute - Visual Functioning Questionnaire (NEI VFQ25) (scores are presented as a number, higher numbers reflect higher QL)

CONTACTS AND LOCATIONS:
Overall Officials: gemma caterina m Rossi, Study Director — IRCCS Fondazione Policlinico San Matteo
Locations (4):
- Italy (4):
  - Dario Sisto, Bari, bari
  - Gemma Caterina Maria Rossi, Pavia, PV
  - Alberto Mavilio, Brindisi
  - Teresa Rolle, Torino

IPD SHARING:
Plan to Share IPD: Yes
data will be published on peer review journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: upon publication
Access Criteria: actually not available